CLINICAL TRIAL: NCT04176497
Title: Image-Adapted Target Volumes Using 68Ga-HBED-CC PSMA-PET/MRI for Unfavorable-Risk Prostate Cancer Patients Receiving Radiation
Brief Title: PSMA-PET/MRI Unfavorable-Risk Target Volume Pilot Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1908
Record Dates: First submitted 2019-11-15; First posted 2019-11-25 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PMSA-PET/MRI (Experimental): Patients scheduled to receive PMSA-PET/MRI scan in addition to standard of care CT scan prior to treatment
  Interventions: Drug: 68Ga-HBED-CC-PSMA

INTERVENTIONS:
Drug: 68Ga-HBED-CC-PSMA — Radioactive tracer used during imaging to help detect PSMA expressing tumor cells.
  Other Names: gallium Ga 68-labeled PSMA-11

SUMMARY:
The goal of this study is to investigate the feasibility and toxicity of using prostate-specific membrane antigen-positron emission tomography (PSMA-PET) and multi-parametric magnetic resonance imagining (mpMRI) with PET-MR technology to define radiotherapy targets, while meeting all the current planning criteria.

DETAILED DESCRIPTION:
PSMA-PET is highly sensitive and specific for detecting prostate cancer. PSMA-PET and mpMRI can potentially help guide target volumes for patients with unfavorable-risk prostate cancer receiving radiation by designing a radiation treatment plan so that the entire prostate receives the prescribed dose of radiation in addition to the visible tumor in the prostate as detected by mpMRI and/or PSMA-PET receiving any inevitable intrinsic plan "hot spots" or areas of dose above the prescription.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Histologically confirmed prostate adenocarcinoma
* Unfavorable intermediate or high-risk, based on the National Comprehensive Cancer Network (NCCN) criteria, with appropriate staging (e.g. bone scan) as defined in the protocol.
* Subject has adequate performance status as defined by ECOG performance status of 0-2.
* Subject is willing and able to comply with the protocol as determined by the Treating Investigator.
* Subject speaks English (quality of life instrument is validated in English).

Exclusion Criteria:

* Contraindications for MRI
* Other prior or concomitant malignancies with the exception of:

  * Non-melanoma skin cancer
  * Other cancer for which the subject has been disease free for ≥5 years before the first study treatment and of low potential risk for recurrence.
* Inflammatory bowel disease
* Absolute contraindications to brachytherapy per American Brachytherapy Society: unacceptable operative risk, absence of rectum, large TURP defects

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male participants only as this is a prostate cancer study
Enrollment: 8 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Repka, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eight subjects were screened, enrolled, and started treatment at one center in the United States between 7/16/2020 and 2/7/2024.
Period: Overall Study
Arm/Group | PMSA-PET/MRI
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who started to study treatment were included.
Arm/Group | PMSA-PET/MRI
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 67.38 [59 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Early Genitourinary and Gastrointestinal Toxicity
Description: Grade 3 or higher early genitourinary and gastrointestinal toxicities, defined by CTCAE version 5.0, include adverse events that develop within three months after starting radiation therapy.
  The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: Up to 22 weeks (3 months after completion of radiation therapy)
Population: Participants started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | PMSA-PET/MRI
Number analyzed (Participants) | 8
Participants | 0

2. Secondary Outcome: Late Genitourinary Toxicity After Radiation
Description: Grade 3 or higher late genitourinary and gastrointestinal toxicities, defined by CTCAE version 5.0, include adverse events that develop three months after starting radiation therapy.
  The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequence
Time Frame: Three months after starting radiation therapy to up to 48 months post-treatment
Population: Participants who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | PMSA-PET/MRI
Number analyzed (Participants) | 8
Participants
  Proctitis (gastrointestinal toxicity) | 1
  Rectal fistula (gastrointestinal toxicity) | 1
  Rectal ulcer (gastrointestinal toxicity) | 1
  Fecal incontinence | 1
  Kidney infection (Pyelonephritis) | 1

3. Secondary Outcome: Biochemical Control Using Prostate-Specific Antigen (PSA) Levels
Description: Biochemical control will be defined according to the Phoenix criteria (PSA rise of <2 ng/mL over nadir). Number of subjects
Time Frame: At 2 years after radiation therapy
Population: We have data available for only 4 subjects at 2 years because of subjects withdrawn, and we do not have 5 years follow-up data for any subjects due to study was terminated by sponsor.
Measure: Count of Participants; unit: Participants
Arm/Group | PMSA-PET/MRI
Number analyzed (Participants) | 4
Participants
  Biochemical control achieved | 4
  Biochemical control not achieved | 0

4. Secondary Outcome: Patient-reported Quality of Life Using Prostate Cancer Symptom Indices (PCSI) Rectal Domain
Description: Patient-reported quality of life in men with prostate cancer can be assessed using the Prostate Cancer Symptom Indices (PCSI), a validated instrument designed to measure disease-specific symptoms and their impact on daily functioning. The PCSI evaluates multiple domains, including urinary function, bowel function, sexual function, and overall well-being. Each domain contains a set of symptom-specific questions rated on a Likert-type scale, typically ranging from 0 (no symptoms or no problem) to 4 or 5 (severe symptoms or major problem). Domain scores were calculated by summing item responses and converting them to a 0-100 scale, where higher scores indicate greater symptom burden.
Time Frame: At 1, 3, 6, 9, 12, 18, 24, 30, 36, 42 months post radiotherapy
Population: Participants started to study intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 1 Month: Data collected at month 1
- 3 Months: Data were collected at 3 moths
- 6 Months: Data collected at 6 months
- 9 Months: Data collected at 9 months
- 12 Months: Data collected at 12 months
- 18 Months: Data collected at 18 months
- 24 Months: Data collected at 24 months
- 30 Months: Data collected at 30 months
- 36 Months: Data collected at 36 months
- 42 Months: Data collected at 42 months
Arm/Group | 1 Month | 3 Months | 6 Months | 9 Months | 12 Months | 18 Months | 24 Months | 30 Months | 36 Months | 42 Months
Number analyzed (Participants) | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 3 | 2 | 1
score on a scale | 98.2 (2.5) | 96.4 (0) | 94 (5.5) | 83.9 (7.6) | 71.4 (15.2) | 96.4 (5.1) | 89.3 (15.2) | 95.2 (8.2) | 100 (0) | 100 (NA) — 1 participant

5. Secondary Outcome: Patient-reported Quality of Life Using Prostate Cancer Symptom Indices (PCSI) - Urinary Domain
Description: as for outcome 4
Time Frame: At 1, 3, 6, 9, 12, 18, 24, 30, 36, 42 months post radiotherapy
Population: Participants started to study intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1 Month | 3 Months | 6 Months | 9 Months | 12 Months | 18 Months | 24 Months | 30 Months | 36 Months | 42 Months
Number analyzed (Participants) | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 3 | 1 | 1
score on a scale | 63.1 (28.7) | 64.4 (8.4) | 68.7 (15.3) | 51.8 (26.2) | 22.6 (6.8) | 53.6 (3.3) | 69.7 (7.7) | 92.9 (9.4) | 78.7 (NA) — 1 participant | 100 (NA) — 1 participant

6. Secondary Outcome: Patient-reported Quality of Life Using the Expanded Prostate Cancer Index Composite (EPIC-26) Bowel Domain
Description: The Expanded Prostate Cancer Index Composite-26 (EPIC-26) is a validated, patient-reported questionnaire designed to assess health-related quality of life among men with prostate cancer. It is a shortened version of the original 50-item EPIC instrument and focuses on five key domains: urinary incontinence, urinary irritation/obstruction, bowel function, sexual function, and hormonal function. EPIC-26 bowel domain reflects symptoms such as bowel urgency, frequency, pain, and overall bowel function. Patients rate each item on a 1-5 scale, and responses are converted to a 0-100 score, with higher scores indicating better bowel function and fewer symptoms. This domain provides a focused measure of how prostate cancer and its treatments affect daily bowel-related quality of life.
Time Frame: At 1, 3, 6, 9, 12, 18, 24, 30, 36, 42 months post radiotherapy
Population: Participants started to study intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 1 Month: Data collected at 1 month
- 3 Months: Data collected at 3 months
Arm/Group | 1 Month | 3 Months | 6 Months | 9 Months | 12 Months | 18 Months | 24 Months | 30 Months | 36 Months | 42 Months
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 1 | 2 | 3 | 2 | 1
score on a scale | 98.6 (2.4) | 95.8 (0) | 86.1 (14.6) | 77.8 (21) | 93.8 (2.9) | 87.5 (NA) — 1 participant | 100 (0) | 88.9 (19.2) | 100 (0) | 100 (NA) — 1 participant

7. Secondary Outcome: Patient-reported Quality of Life Using the Expanded Prostate Cancer Index Composite (EPIC-26) Hormonal Function Domain
Description: The Expanded Prostate Cancer Index Composite-26 (EPIC-26) is a validated, patient-reported questionnaire designed to assess health-related quality of life among men with prostate cancer. It is a shortened version of the original 50-item EPIC instrument and focuses on five key domains: urinary incontinence, urinary irritation/obstruction, bowel function, sexual function, and hormonal function. EPIC-26 hormonal function domain captures symptoms such as fatigue, hot flashes, breast tenderness, and emotional changes. Items are rated on a 1-5 scale and converted to a 0-100 score, with higher scores indicating better hormonal function and fewer symptoms. This domain provides a focused assessment of how prostate cancer and its treatments affect patients' hormone-related quality of life.
Time Frame: At 1, 3, 6, 9, 12, 18, 24, 30, 36, 42 months post radiotherapy
Population: Participants started to study intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1 Month | 3 Months | 6 Months | 9 Months | 12 Months | 18 Months | 24 Months | 30 Months | 36 Months | 42 Months
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 2 | 1 | 2 | 2 | 1 | 1
score on a scale | 70 (28.3) | 57.5 (3.5) | 88.3 (11.5) | 83.3 (16.1) | 95 (7.1) | 62.5 (NA) — 1 participant | 80 (28.3) | 100 (0) | 100 (NA) — 1 participant | 100 (NA) — 1 participant

8. Secondary Outcome: Patient-reported Quality of Life Using the Expanded Prostate Cancer Index Composite (EPIC-26) -Sexual Function Domain
Description: The Expanded Prostate Cancer Index Composite-26 (EPIC-26) is a validated, patient-reported questionnaire designed to assess health-related quality of life among men with prostate cancer. It is a shortened version of the original 50-item EPIC instrument and focuses on five key domains: urinary incontinence, urinary irritation/obstruction, bowel function, sexual function, and hormonal function. EPIC-26 sexual function domain assesses erectile function, ability to achieve orgasm, sexual desire, and overall sexual satisfaction. Items are rated on a 1-5 scale and converted to a 0-100 score, with higher scores reflecting better sexual function and fewer difficulties. This domain provides a focused measure of how prostate cancer and its treatments impact sexual health and related quality of life.
Time Frame: Baseline and at 1, 3, 6, 9, 12, 18, 24, 30, 36, 42 months post radiotherapy
Population: Participants started to study intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1 Month | 3 Months | 6 Months | 9 Months | 12 Months | 18 Months | 24 Months | 30 Months | 36 Months | 42 Months
Number analyzed (Participants) | 1 | 2 | 3 | 3 | 2 | 1 | 2 | 2 | 1 | 1
score on a scale | 43 (NA) — 1 participant | 31.2 (20.6) | 12.2 (10.7) | 8.3 (8.3) | 25.8 (13) | 12.5 (NA) — 1 participant | 36.8 (46.2) | 44 (38.9) | 40.3 (NA) — 1 participant | 69.5 (NA) — 1 participant

9. Secondary Outcome: Patient-reported Quality of Life Using the Expanded Prostate Cancer Index Composite (EPIC-26) Urinary Incontinence, Urinary Irritation Domains
Description: The Expanded Prostate Cancer Index Composite-26 (EPIC-26) is a validated, patient-reported questionnaire designed to assess health-related quality of life among men with prostate cancer. It is a shortened version of the original 50-item EPIC instrument and focuses on five key domains: urinary incontinence, urinary irritation/obstruction, bowel function, sexual function, and hormonal function. EPIC-26 urinary incontinence and urinary irritation/obstruction domains reflects issues such as urine leakage, pad use, urgency, frequency, and weak stream. Items are rated on a 1-5 scale and converted to 0-100 scores, with higher values indicating better urinary function and fewer symptoms. Together, these domains provide a detailed view of how prostate cancer and its treatments affect daily urinary health.
Time Frame: at 1, 3, 6, 9, 12, 18, 24, 30, 36, 42 months post radiotherapy
Population: Participants started to study intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1 Month | 3 Months | 6 Months | 9 Months | 12 Months | 18 Months | 24 Months | 30 Months | 36 Months | 42 Months
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 1 | 2 | 3 | 2 | 1
score on a scale
  Urinary incontinence | 84.8 (13.4) | 76 (33.9) | 82 (13.4) | 63.2 (33.9) | 66.6 (38.4) | 79.2 (NA) — 1 participant | 67.8 (25.1) | 79.2 (36.1) | 92.8 (10.3) | 50 (0)
  urinary irritation | 62.5 (21.7) | 53.1 (13.3) | 89.6 (13) | 77.1 (29.5) | 43.8 (17.7) | 68.8 (NA) — 1 participant | 81.2 (8.8) | 100 (0) | 100 (0) | 100 (0)

10. Secondary Outcome: The Number of Participants Started Study.
Description: The number of participants started study.
Time Frame: Baseline
Population: Participants who screened for the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PMSA-PET/MRI
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: Up to 49 months.
Description: Adverse events were collected from day one of the study treatment to 49 months after completion of treatment. Any hospital admission was graded as a serious adverse event per protocol.
Arm/Group | PMSA-PET/MRI
All-Cause Mortality (participants affected / at risk) | 2/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PMSA-PET/MRI (N=8)
Proctitis (Gastrointestinal disorders) | 1
Rectal ulcer (Gastrointestinal disorders) | 1
Rectal fistula (Gastrointestinal disorders) | 1
Kidney infection (Infections and infestations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PMSA-PET/MRI (N=8)
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 2
Rectal pain (Gastrointestinal disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 7
Urinary retention (Renal and urinary disorders) | 2
Urinary urgency (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Scrotal pain (Reproductive system and breast disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Glaucoma (Eye disorders) | 1
Fatigue (General disorders) | 3
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperlipidemia (Metabolism and nutrition disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 2
Hot flashes (Vascular disorders) | 6
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
This study was terminated before reaching target accrual and follow-up was suspended. Additionally, two versions of the protocol were uploaded since no new participant started to study after amendment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT04176497/Prot_SAP_000.pdf